CLINICAL TRIAL: NCT00859391
Title: A Phase 0 Study in Subjects With Well Controlled Celiac Disease to Assess the Effects of Gluten Digestion With ALV003 (a Protease Enzyme) in Vitro
Brief Title: Effects of Gluten Digestion With ALV003
Acronym: 0801
Status: Completed | Type: Observational
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Dr Gregor Brown, Principal Investigator, Alfred Hospital
Other Study IDs: ALV0801
Record Dates: First submitted 2009-01-19; First posted 2009-03-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Celiac Disease
Keywords: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The enzyme linked immunospot (ELISPOT) assay is used in vaccine development, cancer research, infectious disease diagnosis and monitoring, autoimmune disease studies and allergy and transplantation research. The ELISPOT enables determination of the frequency of cytokine secreting cells. The ELISPOT is a combination of both immunoassay and bioassay because live cells are cultured in plates. This enables a very high sensitivity to detect cytokine secretion at a single cell level as secreted cytokine does not diffuse into media but is immediately membrane bound.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 - Active: This group received gluten pre-treated with ALV003
- 2 - Placebo: This group received Gluten pre-treated with placebo.

SUMMARY:
This is a Phase 0, Double-blind study that will assess the effect of in vitro treatment of gluten with ALV003 or with placebo when ingested by CD Subjects.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effects of gluten treated with ALV003 vs placebo:

* The clinical response by symptom measurement before and after oral challenge
* The immune response measured by ELISPOT testing and serology The secondary objective of the study is to
* Describe the immunotoxic epitope profile of gluten digests with ALV003 compared with placebo

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Well controlled Celiac Disease without flare in symptoms for the past 8 weeks
* History of biopsy proven Celiac Disease
* Able and willing to complete a symptom diary for 3 days prior and through 3 days post gluten challenge
* Been on a gluten free diet for 8 weeks prior to study entry
* Have normal celiac serology (anti- tTG level of <20 units/mL)

Exclusion Criteria:

* Uncontrolled complications of celiac disease which in the opinion of the Investigator would impact their immune response, or pose an increased risk to the subject. (example: like type 1 diabetes or other autoimmune disease)
* Pregnant or breast feeding women, subjects of childbearing potential to use two methods of contraception
* Concomitant medications such as over the counter digestive enzymes, immunosuppressive therapies, anticoagulants, NSAIDs. Chronic medications for well-controlled chronic conditions are allowed.
* Clinically significant abnormal lab values, as determined by the PI:
* Untreated or active peptic ulcer disease, esophagitis, motility disorders or any gastrointestinal diseases.
* Positive pregnancy test within 7 days prior to study drug administration
* Known allergy or hypersensitivity to E.coli or E.coli derived proteins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is patients with celiac disease with HLA DQ2 phenotype who have well controlled celiac disease without significant co-morbidities and are previously on a gluten free diet for at least 8 weeks prior to study entry.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The clinical response by symptom measurement before and after oral challenge | Day 1 and Day 6
The immune response measured by ELISPOT testing and celiac disease serology | Prior to and post 3-day gluten challenge

SECONDARY OUTCOMES:
Describe the immunotoxic epitope profile of gluten digests with ALV003 compared with placebo | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Brown, MD, Principal Investigator — The Alfred
Locations (1):
- Nucleus Networks Limited, Melbourne, Victoria, Australia